CLINICAL TRIAL: NCT02101411
Title: Platelet Reactivity (High On-Treatment Platelet Reactivity) as Guidance for APT (Antiplatelet Therapy) Adjustment After PCI (Percutaneous Coronary Intervention)
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Yueh-Chung, Chen, chief of ICU, Taipei City Hospital
Other Study IDs: TCHIRB-1011207-E-F
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2017-04

CONDITIONS: PRU(Platelet Reactivity Unit); APT(Antiplatelet Therapy); HOTPR(High on Treat Platelet Reactivity)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- clopidogrel: treated with cloopidogrel
  Interventions: Diagnostic Test: PRU(Platelet reactivity unit)
- ticagrelor: treated with ticagrelor
  Interventions: Diagnostic Test: PRU(Platelet reactivity unit)
- cilostazol: treated with clopidogrel+cilostazol
  Interventions: Diagnostic Test: PRU(Platelet reactivity unit)

INTERVENTIONS:
Diagnostic Test: PRU(Platelet reactivity unit) — measure by VeryfyNow.
  Other Names: Platelet reactivity unit

SUMMARY:
Since thrombus formation is a very complex procedure in vivo, platelet function testing methods in vitro might only reflect the degree of inhibition of platelet from a certain level, which do't reflect the functional status of platelets in vivo adequately. There are a variety of signal transduction pathways involved in the formation of platelet activation and thrombosis. Gurbel et al. first reported individuals with variability on clopidogrel treatment response in 2003, and proposed the concept of clopidogrel resistance. Different patients received the same dose of aspirin or other anti -platelet drug such as clopidogrel , due to various reasons bound to lack some patients antithrombotic efforts to increase the incidence of thrombotic events , while another part of the patient easily understood antithrombotic excessive bleeding events, " antithrombotic individualized treatment , " according to differences in patient against platelet drugs or anticoagulant drug reactions and adjust the treatment plan , is the direction of antithrombotic therapy in the future.

There are a number of studies have shown that patients with no response Clopidogrel , measuring the relationship between high platelet reactivity and clinical adverse ischemic events displayed between platelet activity . However, there is still lack of quantitative threshold high platelet reactivity and the risks associated with the clinical consensus . In addition, there are only limited data support, to measure platelet function -based therapy to improve the clinical efficacy of the concept . Over the years, more than 20,000 cases reported in patients with numerous studies confirm that high platelet reactivity after PCI with stent thrombosis , including cardiovascular events , including an increased risk of significant correlation . Pharmacodynamic analysis GRVITAS trial showed significantly lower platelet reactivity associated with a lower risk of adverse cardiovascular events . Brar in more than 3000 cases of patients published in JACC Meta-analysis showed that "high platelet reactivity " of patients whose cardiovascular death, heart attack and stent thrombosis occurred more than twice the rate of " non-high platelet reactivity " patients .

Two new anti-platelet drugs (Prasugrel and Ticagrelor) in several recent randomized trials have considerable persuasive , and has included some guidance in the current guidelines. Ticagrelor even more than Prasugrel in pharmacodynamic studies more effectively inhibit platelet , and has a lower risk of bleeding. Cilostazol is an old drug , mostly for the treatment of intermittent claudication , in recent years there are also some testing and coronary stents prevent restenosis after angioplasty , however, so far , there is little direct comparison Cilostazol and Ticagrelor related articles .

We designed this test , in addition to testing for high yellow people treat DAPT (dual anti-platelet therapy) under the platelet reactivity (high on-treatment platelet reactivity) ratio , this population of patients with ticagrelor instead for a month or cilostazol treatment after its platelet reactivity changes and compare between the two groups , and even track six months after the bleeding and adverse cardiovascular events rate? Through this test we can compare the treatment for patients with high platelet reactivity of what strategies more appropriate.

ELIGIBILITY:
Inclusion Criteria:

1 under DAPT (dual antiplatelet therapy) of stable angina patients for elective stent implantation.

2. DAPT 24 hours, 7d and 30d after treatment PRU (platelet activity units) values. (Drug unresponsive patients was defined as PRU> 235).

Exclusion Criteria:

1.Not suitable for the treatment of patients with DAPT. (Active peptic ulceration or bleeding) 2 patients of aspirin, clopidogrel, ticagrelor, cilostazol medication intolerance.

3 contraindications for aspirin, clopidogrel, ticagrelor, cilostazol drug usage (such as heart failure patients not suitable for use cilostazol).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stable angina who received routine dual antiplatelet agents therapy.
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yueh Chung, chief doctor, Study Chair — taipei city hospital, taipei city goverment; Chen Yueh Chung, chief doctor, Study Chair — taipei city hospital, tiapei city goverment
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen YC, Lin FY, Lin YW, Cheng SM, Lin RH, Chuang CL, Sheu JS, Chen SM, Chang CC, Tsai CS. DAPT Plus Cilostazol is Better Than Traditional DAPT or Aspirin Plus Ticagrelor as Elective PCI for Intermediate-to-Highly Complex Cases: Prospective, Randomized, PRU-Based Study in Taiwan. Am J Cardiovasc Drugs. 2019 Feb;19(1):75-86. doi: 10.1007/s40256-018-0302-3. PMID 30467686

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin+Clopidogrel: aspirin 100mg qd+clopidogrel 75mg qd
- Aspirin+Ticagrelor: aspirin100mg qd+ticagrelor 90mg bid
- Aspirin+Clopidogrel+Cilostazol: aspirin 100mg qd+clopidogrel 75mg qd+cilostazol 100mg bid
Period: Overall Study
Arm/Group | Aspirin+Clopidogrel | Aspirin+Ticagrelor | Aspirin+Clopidogrel+Cilostazol
Started | 111 | 109 | 114
Completed | 107 | 102 | 104
Not Completed | 4 | 7 | 10

BASELINE CHARACTERISTICS:
Population: PRU after anti-platelet drugs
Groups:
- Aspirin+Clopidogrel; Aspirin+Clopidogrel+Cilostazol: aspirin 100mg qd+clopidogrel 75mg q...
- Total: Total of all reporting groups
Arm/Group | Aspirin+Clopidogrel | Aspirin+Ticagrelor | Aspirin+Clopidogrel+Cilostazol | Total
Number analyzed (Participants) | 107 | 102 | 104 | 313
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 86 | 83 | 80 | 249
  >=65 years | 21 | 19 | 24 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (13) | 66.1 (13.9) | 65.2 (13.4) | 65.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 29 | 24 | 86
  Male | 74 | 73 | 80 | 227
Region of Enrollment [Number; unit: participants]
  Taiwan | 107 | 102 | 104 | 313

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants With MACE(Major Adverse Cardiac Event) of Study Subjects
Description: MACE(major adverse cardiac event) include: death, myocardial infarction, revascularization.
Time Frame: 24 months
Measure: Number; unit: numbers of participants with MACE
Arm/Group | Aspirin+Clopidogrel | Aspirin+Ticagrelor | Aspirin+Clopidogrel+Cilostazol
Number analyzed (Participants) | 107 | 102 | 104
numbers of participants with MACE | 1 | 1 | 2
Statistical Analysis 1: Comparison: Aspirin+Clopidogrel vs Aspirin+Ticagrelor vs Aspirin+Clopidogrel+Cilostazol; The differences among the three PRU groups (<85, 85-208,>208) and MACE rate at 24 months were compared using the Chi-squared test. was recorded; Test type: Other — The Chi-squared test was used for comparisons of all categorical variables. If 20% of the cells had an expected value < 5, then Fisher's exact test was used; p = 0.002, Chi-squared — The Chi-squared test was used for comparisons of all categorical variables. If 20% of the cells had an expected value < 5, then Fisher's exact test was used; The differences among the three PRU groups (<85, 85-208,>208) and ADEs were compared using the Chi-squared test; Hazard Ratio (HR) = 1.19, Standard Deviation 0.005
Statistical Analysis 2: Comparison: Aspirin+Clopidogrel vs Aspirin+Ticagrelor vs Aspirin+Clopidogrel+Cilostazol; The differences among the three PRU groups (<85, 85-208,>208) and ADEs were compared using the Chi-squared test; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.002, Chi-squared — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, Standard Deviation 0.005

ADVERSE EVENTS:
Time Frame: 24m
Arm/Group | Aspirin+Clopidogrel | Aspirin+Ticagrelor | Aspirin+Clopidogrel+Cilostazol
All-Cause Mortality (participants affected / at risk) | 1/107 | 1/102 | 2/104
Serious Adverse Events (participants affected / at risk) | 1/107 | 0/102 | 2/104
Other Adverse Events (participants affected / at risk) | 0/107 | 0/102 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin+Clopidogrel (N=107) | Aspirin+Ticagrelor (N=102) | Aspirin+Clopidogrel+Cilostazol (N=104)
1 (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) — Myocardial infarction, or related death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No